CLINICAL TRIAL: NCT06291467
Title: Plasma Beta-endorphin Levels and Suicidal Behavior
Acronym: BEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Institut de Génomique Fonctionnelle (IGF) de Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL23_0121
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-01

CONDITIONS: Suicide; Depression; Beta Endorphin
Keywords: suicide; depression; beta endorphin
MeSH Terms: conditions — Suicide; Depression | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suicide attempters (Experimental): patients hospitalized for suicide attempt within the last 72 hours
  Interventions: Biological: Blood samples; Other: questionnaires
- Affective controls (Active Comparator): patients hospitalized for current major depressive episode according to DSM-5 criteria and without any lifetime history of suicide attempt
  Interventions: Biological: Blood samples; Other: questionnaires

INTERVENTIONS:
Biological: Blood samples — Blood samples will be collected at both visit between 8:30 a.m. and 9:30 a.m. and fasting from midnight.
Other: questionnaires — Questionnaires will be administrated at both visits to assess the suicide spectrum, the depression level and some personality traits.
  Hetero-questionnaires will be administrated during a clinical interview conducted by a psychiatrist or psychologist at the inclusion.
  * MINI 7.0 Mini-International Neuropsychiatric Interview :
  * MADRS (Montgomery Asberg Depression Scale)
  * C-SSRS (Columbia-Suicide Severity Rating Scale)
  * FAST (Functioning Assessment Short Test)
  Self-administered questionnaire will be completed by the participant at the inclusion and at the end of hospitalisation (D7+/- 2 days) :
  * STAI-Y (State-Trait Anxiety Inventory )
  * PPP-VAS (Visual Analog Scale to measure Psychological and Physical Pain)
  * SHAPS (Snaith-Hamilton-Pleasure Scale )
  * CTQ (Childhood Trauma Questionnaire)
  * ESUL : Echelle de solitude de l'université de Laval
  * BIS-11 : (Barratt Impulsiveness Scale)
  * QIDS (Quick Inventory of Depressive Symptomatology)

SUMMARY:
It is an interventional research, monocentric, which involves only minimal risks and constraints.

Psychological pain is closely associated with suicidal ideation (SI) and suicidal behavior, regardless of the severity of the depression. The psychological pain being regulated by the opioidergic system, it seems that a dysfunction of this system exists in suicidal attempters. The aim of this study is to explore the association between levels of β-endorphin and suicidal behavior.

The research team will measure plasma levels of β-endorphin in patients hospitalized for suicide attempt (SA) within 72 hours and compare them to those of patients hospitalized for current major depressive episode (EDC) without any lifetime history of SA. In order to follow the kinetics of β endorphin levels, The research team will carry out two measurements: at inclusion and on day 7 (+/- 2 days) of inclusion.

The main objective is to compare plasma β-endorphin levels in patients hospitalized following a recent SA (≤72 hours) and in patients hospitalized for an EDC without lifetime history of SA.

DETAILED DESCRIPTION:
104 participants will be enrolled, divided into 2 groups:

group 1: 52 Suicide attempters, currently hospitalized patients for a suicide attempt within the 72 last hours group 2: 50 Affective controls, currently hospitalized patients for current major depressive episode according to the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria and without any lifetime history of suicide attempt;

The protocol includes two visits.The first visit is the inclusion visit carried out at the beginning of patient hospitalization, within 72 hours following suicide attempt (SA) for group 1 (suicide attempters) and within 72 hours following the admission to hospital for group 2 (affective controls).

The second visit takes place at the end of hospitalisation, on Day 7 +/- 2 days, after SA for group 1 and after admission to hospital for group 2 .

At each visit, a clinical assessment will be performed to characterise psychopathology and suicidal characteristics. Blood samples will be obtained in order to measure beta-β-endorphin levels.

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criteria:
* Aged between 18 and 65 years old,
* Subject with a psychiatric diagnosis of current major depressive episode according to DSM-5 criteria
* Able to understand the nature, purpose and methodology of the study

Specific inclusion criteria

* Suicide attempters: Subject hospitalized for of proven suicide attempt (<72h)
* Affective controls: Subject hospitalized for a current major depressive episode according to DSM-5 criteria and without any lifetime history of suicidal behavior (proven, interrupted or aborted)

Non inclusion criteria

* Diagnosis of bipolar disorder
* Lifetime diagnosis of schizoaffective disorder, schizophrenia or unspecified psychosis
* Current diagnostic of illicit substance / alcohol use disorder within the last 6 months
* Diabetes or obesity (BMI > 29)
* Inflammatory disease (e.g. Lupus, Rheumatoid Arthritis)
* Receiving opiate treatment or opiate substitution treatment
* Law protected ( guardianship or curatorship)
* Deprived of liberty (by judicial or administrative decision or forced hospitalization)
* Pregnant and breastfeeding women
* Inability to understand, speak and write French
* Refusal to participate in the study.
* Not be affiliated to a French National Social Security System

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Comparison of plasma β-endorphin levels between patients with recent suicide attempt (≤ 72 hours) vs. patients with current major depressive episode without any lifetime history of suicide attempt. | Baseline and day 7± 2 days
  blood sample between 8:30 a.m. and 9:30 a.m for β-endorphin dosage (pg/mL)

SECONDARY OUTCOMES:
- The kinetics of β-endorphin levels between two measurement points (inclusion and D7+/-2 days) in patients with recent suicide attempt (≤ 72 hours) vs. patients with current major depressive episode without any history of suicide attempt. | Baseline and day 7± 2 days
  blood sample between 8:30 a.m. and 9:30 a.m for β-endorphin dosage (pg/mL)
The level of depression in the last week before inclusion assessed by a self-administered questionnaire (MADRS) | Baseline and day 7± 2 days
  MADRS (Montgomery and Asberg Depression Rating Scale, hetero-assessment) is a 10-item questionnaire with a score ranging from 0 to 60 (the higher the score, the more depressive symptoms are present) .
The level of depression in the last week before inclusion assessed by a self-administered questionnaire (QIDS-16) | Baseline and day 7± 2 days
  the QIDS-16 (Quick Inventory of Depressive Symptomatology, self-questionnaire) is a 16 items questionnaire, scored from 0 to 3,The total score ranges from 0 (no depression) to 42 (severe depression).
To assess the association between β-endorphin levels and and Suicidal ideation and history of suicidal behavior in the last week before inclusion, | Baseline and day 7± 2 days
  Assessed with the CSSRS (Columbia Suicide Severity Rating Scale, hetero-assessment) questionnaire used for suicide assessment with a scale from 0 to 5 (highest suicidal risk)
To assess the association between β-endorphin levels and Anhedonia | Baseline and day 7± 2 days
  assessed with the SHAPS (Snaith and Hamilton pleasure scale, self-assessment)14 items scoring 0 to 3 for each item (the lower the score, the lower the pleasure)
To assess the association between β-endorphin levels and Current psychological and physical pain as well as usual and maximum over the 15 days before inclusion | Baseline and day 7± 2 days
  assessed with a numerical scale (Visual Analog Scale to measure Psychological and Physical Pain : PPP-VAS, self-questionnaire scoring 0 to 10, the lower the score, the less pain.
To assess the association between β-endorphin levels and Anxiety, | Baseline and day 7± 2 days
  Assessed with the STAI (trait and state anxiety assessment scale, self-questionnaire) composed of 2 distinctive scale. Each consists of 20 items rated from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte NOBILE, Pharm D, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No